CLINICAL TRIAL: NCT00589459
Title: A Pilot Study of Gender Differences in the Prevalence of Undiagnosed Diabetes in Acute Coronary Syndromes (ACS)
Brief Title: Gender Differences in Prevalence of Undiagnosed Diabetes in ACS
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other); Ethel F Donaghue Women's Health Investigator's Program at Yale (Unknown)
Responsible Party: Barbara I Gulanski, MD, MPH, Yale University School of Medicine
Other Study IDs: 12258; AHA; Donaghue Women's Health R02524
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pre-diabetes; Diabetes
Keywords: undiagnosed diabetes; undiagnosed pre-diabetes; acute coronary syndrome; undiagnosed pre-diabetes and undiagnosed diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: non-diabetic women with acute coronary syndrome (ACS)
- 2: non-diabetic men with acute coronary syndrome (ACS)

SUMMARY:
The primary goal of this study is to measure the prevalence of undiagnosed pre-diabetes/diabetes among women hospitalized with acute coronary syndromes (ACS) compared to men. Inpatients with confirmed ACS (and no known prior history of diabetes) are invited to return to the Yale Hospital Research Unit 6-8 weeks after hospital discharge for an oral glucose tolerance test to identify individuals with pre-diabetes and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome
* age > 30 yrs

Exclusion Criteria:

* previously diagnosed diabetes
* ACS due to substance abuse or trauma

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men admitted with an acute coronary syndrome who do not have a prior diagnosis of diabetes
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2001-10-01 (Actual); Primary Completion 2005-09-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of undiagnosed pre-diabetes or undiagnosed diabetes | after hospitalization for acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Gulanski, MD, MPH, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale Center for Clinical Investigation, New Haven, Connecticut